CLINICAL TRIAL: NCT01143896
Title: Hepatitis C Translating Initiatives for Depression Into Solutions
Brief Title: Hepatitis C Translating Initiatives for Depression Into Effective Solutions
Acronym: HEPTIDES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SDP 10-044; 10-05 (Other: VA Central IRB)
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Results first posted 2016-04-11 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Hepatitis C; Depression
Keywords: Hepatitis C; Depression; Collaborative care; Antiviral treatment
MeSH Terms: conditions — Hepatitis C; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Depression Collaborative Care (Experimental): Depression collaborative care: includes a stepped-care model. The 5 steps include symptom and self-management monitoring by a depression care manager (DCM) and the following: 1) watchful waiting, 2) treatment recommendations (counseling or pharmacotherapy), 3) pharmacotherapy recommended by a Clinical Pharmacist, 4) combination pharmacotherapy and specialty mental health counseling, and 5) referral to mental health. The DCM: provides education about depression and depression treatment options; assesses the patient's treatment preferences and barriers, and the patient's current depression severity and mental health comorbidity; initiates a patient self-management plan, and assess treatment adherence. The DCM uses standard alcohol screening and brief intervention. The DCM also screens for street drug use and recommends referral for to the local substance abuse treatment programs.
  Interventions: Other: Depression collaborative care model
- Arm 2: Usual Care (No Intervention): Usual care will include depression screening with the same PHQ-9 screener used for Arm 1. The depression collaborative care team will not be a part of the usual care condition.

INTERVENTIONS:
Other: Depression collaborative care model — The intervention will include a stepped-care model. The 5 steps include symptom and self-management monitoring by a depression care manager (DCM) and the following: 1) watchful waiting, 2) treatment recommendations (counseling or pharmacotherapy), 3) pharmacotherapy recommended by a Clinical Pharmacist, 4) combination pharmacotherapy and specialty mental health counseling, and 5) referral to mental health. The DCM: provides education about depression and depression treatment options; assesses the patient's treatment preferences and barriers, and the patient's current depression severity and mental health comorbidity; initiates a patient self-management plan, and assess treatment adherence. The DCM uses standard alcohol screening and brief intervention. The DCM also screens for street drug use and recommends referral for to the local substance abuse treatment programs.
  Arms: Arm 1: Depression Collaborative Care

SUMMARY:
Chronic infection with hepatitis C (CHC) is a common and expensive condition, and it disproportionately affects Veterans. Treatment with antiviral therapy reduces liver disease progression and improves health related quality of life. However, ~70% of Veterans with CHC are considered ineligible for antiviral treatment. Most of these patients are excluded due to the presence of co-existing depression and substance use. The proposed project will adapt and adopt an evidence-based collaborative depression care model in CHC clinics. By removing the leading contraindication for antiviral treatment, this project will potentially yield benefits that go far beyond the obvious quality of life benefit from antidepressant therapy itself.

DETAILED DESCRIPTION:
Project Background and Rationale: Depression is highly prevalent, yet under-diagnosed and under-treated in CHC. Treatment models that increase collaborative management of depression by mental health and physical health clinicians can improve quality and outcomes, and collaborative care models have been identified as the best-practice for depression in VA primary care settings. However, the antiviral treatment for CHC patients may not benefit from the existing primary care-mental health integration because the antiviral treatment is time-limited and conducted in specialty clinics. Although there is little evidence evaluating the effects of collaborative depression care in specialty settings, QUERI HIV-hepatitis initiated one of the first such efforts that effectively implemented collaborative depression care in HIV clinics. Built on this experience, an intensive yet focused collaborative care model in CHC clinics may be effective in improving not only depression but also CHC care. This proposed study, "Hepatitis-Translating Initiatives for Depression into Effective Solutions (HEP-TIDES)" will target this issue.

Project Objectives: The proposal has three overarching primary aims and one exploratory aim. The primary aims are (1) adapt and adopt the collaborative care model for improving depression care in specialty CHC care settings, (2) compare the effectiveness of HEP-TIDES to usual care in improving CHC care, and (3) compare the effectiveness of HEP-TIDES to usual care in improving depression care. The exploratory aim is to evaluate the cost-effectiveness of HEP-TIDES versus usual care.

Project Methods: HEP-TIDES is a multi-site, multi-method implementation project. HEP-TIDES will use evidence-based quality improvement (EBQI) methods to adapt and implement depression screening and the collaborative care model for depression in the CHC clinics at 4 disparate VA facilities (aim 1). HEP-TIDES will involve CHC and mental health providers working with an off-site depression care team comprised of a depression care nurse manager, pharmacist, and a psychiatrist. The purpose of the team will be to support CHC and mental health clinicians in delivering evidence-based stepped-care depression treatment. The adapted model will also take into account the substance use disorders among CHC patients. HEP-TIDES implementation will be assessed using a formative evaluation of the implementation process and a summative evaluation of a randomized controlled implementation trial of collaborative depression care in 242 patients (aims 2 and 3).

ELIGIBILITY:
Inclusion Criteria:

* confirmed untreated infection (positive HCV RNA test)
* current PHQ-9 score of 10 or more
* current treatment in the CHC clinic

Exclusion Criteria:

* non-Veterans
* patients who do not have access to a telephone
* patients with current suicidal ideation
* patients with significant cognitive impairment as indicated by a score > 10 on the Blessed Orientation Memory and Concentration Test
* patients with a chart diagnosis of schizophrenia
* patients with a chart diagnosis of bipolar disorder who have been hospitalized for a mental health condition within the last 12 months

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2012-02; Primary Completion 2014-09 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fasiha Kanwal, MBBS MD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX; Jeffrey M. Pyne, MD, Principal Investigator — Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR; Brian Dieckgraefe, MD, Principal Investigator — St. Louis VA Medical Center John Cochran Division, St. Louis, MO; Matthew Goetz, MD, Principal Investigator — VA Greater Los Angeles Healthcare System
Locations (4):
- United States (4):
  - Central Arkansas VHS Eugene J. Towbin Healthcare Ctr, Little Rock, Little Rock, Arkansas
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - St. Louis VA Medical Center John Cochran Division, St. Louis, MO, St Louis, Missouri
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas

REFERENCES:
- [Result] Pyne JM. Expanding the Scope of Integrated Behavioral Health Care for Patients With Hepatitis C Virus. Clin Gastroenterol Hepatol. 2015 Nov;13(11):2015-6. doi: 10.1016/j.cgh.2015.04.174. Epub 2015 May 5. No abstract available. PMID 25952310
- [Result] Zuchowski JL, Hamilton AB, Pyne JM, Clark JA, Naik AD, Smith DL, Kanwal F. Qualitative analysis of patient-centered decision attributes associated with initiating hepatitis C treatment. BMC Gastroenterol. 2015 Oct 1;15:124. doi: 10.1186/s12876-015-0356-5. PMID 26429337
- [Derived] Kanwal F, Pyne JM, Tavakoli-Tabasi S, Nicholson S, Dieckgraefe B, Storay E, Bidwell Goetz M, Smith DL, Sansgiry S, Gifford A, Asch SM. Collaborative Care for Depression in Chronic Hepatitis C Clinics. Psychiatr Serv. 2016 Oct 1;67(10):1076-1082. doi: 10.1176/appi.ps.201400474. Epub 2016 Jul 1. PMID 27364808

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited a total of 309 patients from CHC clinics at 4 VAs (Houston, St Louis, Little Rock, and Los Angeles) between April 2012 and September 2013. Of these, 292 patients completed baseline interviews. Follow-up data-collection interviews were completed for 263 (90.1%) participants at 6-months and 242 (78.3%) participants at 12-months.
Groups:
- Arm 1: Depression Collaborative Care: Depression collaborative care model: The depression collaborative care arm will include a stepped-care model. The five steps are expected to include symptom and self-management monitoring by depression care manager (DCM) and the following: 1) watchful waiting, 2) treatment recommendations (counseling or pharmacotherapy), 3) pharmacotherapy recommended by a Clinical Pharmacist, 4) combination pharmacotherapy and specialty mental health counseling, and 5) referral to mental health. The DCM will provide education about depression and depression treatment options, assess the patient's treatment preferences and barriers, assess the patient's current depression severity and mental health comorbidity, initiate a self-management plan, and assess treatment adherence. The DCM will use the alcohol screening and brief intervention. The DCM will also screen for street drug use and will recommend referral of participants who are using street drugs to the local substance abuse treatment programs.
Period: Overall Study
Arm/Group | Arm 1: Depression Collaborative Care | Arm 2: Usual Care
Started | 156 | 153
Completed | 114 | 128
Not Completed | 42 | 25
Not completed — Did not complete Baseline Interview | 5 | 4
Not completed — Lost to Follow-up | 18 | 13
Not completed — Withdrawal by Subject | 13 | 5
Not completed — Death | 6 | 3

BASELINE CHARACTERISTICS:
Population: A total of 292 participants completed baseline interviews.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Depression Collaborative Care | Arm 2: Usual Care | Total
Number analyzed (Participants) | 145 | 147 | 292
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (5.8) | 59 (5.2) | 59 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 139 | 141 | 280
Race/Ethnicity, Customized [Number; unit: participants]
  White Non-Hispanic | 59 | 41 | 100
  Black or African American | 72 | 91 | 163
  Other | 14 | 15 | 29
Region of Enrollment [Number; unit: participants]
  United States | 145 | 147 | 292
Marital Status [Number; unit: participants]
  Single, Never Married | 45 | 68 | 113
  Married | 14 | 16 | 30
  Other (divorced, widowed, separated, no response) | 86 | 63 | 149
Annual Income [Number; unit: participants]
  Less than $20,000 | 60 | 57 | 117
  Over $20,000 | 43 | 41 | 84
  Don't Know/Refused | 42 | 49 | 91
History of Mood Disorders [Number; unit: participants] — In the last 6 months, did you receive care for personal or emotional problems, feeling down, worried or anxious, or alcohol or drug problem?
  participants
    Yes | 65 | 67 | 132
    No | 80 | 78 | 158
    Don't Know/Refused | 0 | 2 | 2
Taking antidepressant meds at baseline [Number; unit: participants] — Do you have a current prescription for any anti-depressant medications, such as prozac or lexapro?
  participants
    Yes | 71 | 67 | 138
    No | 71 | 79 | 150
    Don't Know/Refused | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Initiated Hepatitis C Antiviral Treatment Within 12 Months of Enrollment
Description: Antiviral treatment initiation was measured dichotomously by assigning a value of 1 if the patient received at least one prescription of interferon within 12 months of enrollment, and a value of 0 otherwise.
Time Frame: 12 months
Population: intent to treat
Measure: Number; unit: participants
Arm/Group | Arm 1: Depression Collaborative Care | Arm 2: Usual Care
Number analyzed (Participants) | 114 | 128
participants | 11 | 7

2. Secondary Outcome: Quality of Hepatitis C Care: Quality Indicators: Proportion of QIs Received
Description: Quality of CHC Indicator Measure is based on a Delphi panel-derived list of quality indicators (QI) in CHC care. The list spans the following domains of care, i.e., CHC-specific function of care (diagnosis, specialty evaluation, treatment, etc); general function of care (diagnosis, treatment, follow-up); and mode of care (encounter, medication, immunization, counseling, etc). Adherence to a given QI is scored as 1 if there is evidence in the patient EMR for the indicator being satisfied. The quality of CHC care at the patient level is calculated by dividing the number of QIs for which that individual received the indicated care by the number of QIs for which the individual is eligible for during the length of time the patient is enrolled in the HEP-TIDES 12-month study timeframe.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: proportion of QIs met
Arm/Group | Arm 1: Depression Collaborative Care | Arm 2: Usual Care
Number analyzed (Participants) | 114 | 128
proportion of QIs met | .89 (.16) | .83 (.19)

3. Secondary Outcome: Medication Adherence: Medication Possession Ratio
Description: Medication adherence was measured using the Medication Possession Ratio (MPR) calculation: Pharmacy refill data was used to calculate a medication possession ratio (MPR), by dividing the number of days supply of a medication received by the number of day's supply the patient needed to be able to take the medication continuously. An MPR closer to 1.0 indicates better adherence and has been associated with lower rates of hospital admission in veterans and greater symptom improvement.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: medication posession ratio
Arm/Group | Arm 1: Depression Collaborative Care | Arm 2: Usual Care
Number analyzed (Participants) | 114 | 128
medication posession ratio | .83 (.20) | .78 (.24)

4. Primary Outcome: Depression Care: Treatment Response
Description: Depression outcomes were assessed using the item mean score from the 20-item Hopkins Symptom Checklist (SCL-20) collected at baseline and 12-months. The SLC-20 items are scored from 0 to 4 and averaged to provide a mean depression severity score ranging from 0 to 4. Depression treatment response was defined as a 50% or greater decrease in the mean SCL-20 score compared with baseline.
Time Frame: Baseline and 12 months
Measure: Number; unit: participants
Arm/Group | Arm 1: Depression Collaborative Care | Arm 2: Usual Care
Number analyzed (Participants) | 114 | 128
participants | 36 | 19

5. Primary Outcome: Depression Care: Depression Remission
Description: Depression outcomes were assessed using the item mean score from the 20-item Hopkins Symptom Checklist (SCL-20) collected at baseline and 12-months. The SLC-20 items are scored from 0 to 4 and averaged to provide a mean depression severity score ranging from 0 to 4. Remission was defined as an item mean SCL-20 score of less than 0.5.
Time Frame: Baseline and 12 months
Measure: Number; unit: participants
Arm/Group | Arm 1: Depression Collaborative Care | Arm 2: Usual Care
Number analyzed (Participants) | 114 | 128
participants | 22 | 9

6. Primary Outcome: Depression Care: Change From Baseline in Number of Depression Free Days (DFDs) at 12 Months
Description: The change in Depression Free Days was assessed using the item mean score from the 20-item Hopkins Symptom Checklist (SCL-20) collected at baseline and 12-months. The SLC-20 items are scored from 0 to 4 and averaged to provide a mean depression severity score ranging from 0 to 4. Depression-free days (DFDs) were calculated using an SCL-20 score of less than 0.5 for depression-free and 2.0 or higher for fully symptomatic, and scores in between were assigned a linear proportional value.
Time Frame: From Baseline to 12 months
Measure: Mean (Standard Deviation); unit: Depression Free Days (DFDs)
Arm/Group | Arm 1: Depression Collaborative Care | Arm 2: Usual Care
Number analyzed (Participants) | 114 | 128
Depression Free Days (DFDs) | 118.74 (106.68) | 109.30 (117.88)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Arm 1: Depression Collaborative Care | Arm 2: Usual Care
Serious Adverse Events (participants affected / at risk) | 6/145 | 3/147
Other Adverse Events (participants affected / at risk) | 0/145 | 0/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Depression Collaborative Care (N=145) | Arm 2: Usual Care (N=147)
Death (IRB determined unrelated to the study) (General disorders) | 6 (6) | 3 (3) — Specific cause of death unavailable

LIMITATIONS AND CAVEATS:
Primary Outcome Initiation of HCV treatment was affected by the 2012 announcement that new interferon-sparing antiviral drugs might be released within 1 year. Most HCV clinicians advised patients to wait for the new drugs (released in 2014).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes